CLINICAL TRIAL: NCT07196358
Title: ROLE OF HEPARIN TO PREVENT HYPERTROPHIC SCARNIG IN DONOR AREA OF SPLIT THICKNESS SKIN GRAFT
Brief Title: Topical Heparin for Prevention of Hypertrophic Scarring in Split-Thickness Skin Graft Donor Sites
Acronym: HepScar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Ruth K.M. Pfau Civil Hospital, Karachi (Other Government)
Responsible Party: Principal Investigator, Asma Ishtiaq, DR, Dr. Ruth K.M. Pfau Civil Hospital, Karachi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: DUHS-185; IRB-3459-DUHS/Approval-2024-18 (Other: DUHS)
Record Dates: First submitted 2025-09-21; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hypertrophic Scarring; Pain, Postoperative; Wound Healing
Keywords: Hypertrophic Scar Split-Thickness Skin Graft (STSG) Donor Site Wound Healing Topical Heparin Scar Prevention Vancouver Scar Scale Pain Management
MeSH Terms: conditions — Cicatrix, Hypertrophic; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: This is an open-label, parallel-group randomized controlled trial. Participants will act as their own controls, with one thigh receiving a heparin-soaked dressing (intervention) and the other thigh receiving the standard dressing (control). This design allows for direct comparison of hypertrophic scarring and pain outcomes at donor sites under different dressing protocols while controlling for individual patient variability. The intervention will be applied immediately after split-thickness skin graft harvesting and maintained according to the study protocol.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1: Standard Dressing (Active Comparator): Description: Donor site of STSG treated with standard dressing (paraffin gauze, gauze pieces, bandaged) as per hospital protocol. Dressing removed on 10th post-operative day unless clinically indicated earlier.
  Interventions: Other: Standard dressing
- Heparin Dressing (Experimental): Description: Donor site of STSG treated with heparin-soaked gauze (5 ml 5000 IU/ml heparin diluted in 50 ml saline to 500 IU/ml concentration) applied immediately post-harvest, dressing left in place till 10th post-operative day unless clinically indicated earlier.
  Interventions: Other: Topical Heparin Dressing

INTERVENTIONS:
Other: Standard dressing — Intervention Description: Donor site of STSG treated with standard dressing. Wound is cleaned, paraffin gauze applied, covered with gauze pieces and bandaged. Dressing is removed on the 10th post-operative day, or earlier if excessive exudate is present. Pain and wound healing monitored per standard care protoco
  Arms: Arm 1: Standard Dressing
Other: Topical Heparin Dressing — Intervention Description: Donor site of STSG treated with heparin dressing. 5 ml of 5000 IU/ml heparin is diluted in 50 ml normal saline to produce 500 IU/ml concentration. Gauze is soaked in this solution and applied to donor site immediately after graft harvest. Dressing remains in place until 10th post-operative day unless clinical indication requires earlier change. Pain, wound healing, and hypertrophic scarring assessed during follow-up.
  Arms: Heparin Dressing

SUMMARY:
This study is testing whether applying a special dressing soaked with heparin (a medicine that improves blood flow and reduces scar formation) can help prevent thick, raised scars (called hypertrophic scars) and reduce pain at the site where skin is taken for a split-thickness skin graft. When people need skin grafts for burns, injuries, or other conditions, the area where the skin is taken (donor site) can sometimes heal with painful or raised scars. In this study, each patient will have one donor site treated with the standard dressing and the other site treated with heparin dressing. We will compare how the wounds heal, the amount of pain, and whether scars develop over a 3-month period. The goal is to see if this simple, low-cost method can improve healing and reduce scarring for patients needing skin grafts.

DETAILED DESCRIPTION:
Hypertrophic scarring at the donor site of split-thickness skin grafts (STSG) is a common problem that can cause pain, itching, discomfort, and cosmetic concerns. Conventional donor site dressings allow healing but do not specifically address scar prevention. Heparin has anti-inflammatory and anti-fibrotic properties, improves local blood circulation, and may reduce the formation of raised scars. Previous research has suggested a role for topical heparin in burn wound management, but its effect on STSG donor sites has not been adequately studied.

This study is an open-label, randomized controlled trial conducted in the Plastic & Reconstructive Surgery Department at Ruth Pfau Civil Hospital, Dow University of Health Sciences. A total of 200 patients requiring STSG will be enrolled. Each patient will provide two donor sites (both thighs). One site will receive the standard paraffin gauze dressing, while the other will receive a heparin-soaked gauze dressing prepared by diluting heparin 5000 IU/mL with saline to achieve a 500 IU/mL solution. Dressings will remain in place until postoperative day 10 unless earlier change is required.

The primary outcome is the incidence and severity of hypertrophic scarring at the donor site, assessed using the Vancouver Scar Scale at 3 months. Secondary outcomes include donor site pain (measured by Numeric Rating Scale), analgesic requirements, and wound complications. Patients will be followed up at day 10, 1 month, and 3 months.

The study aims to determine whether topical heparin is an inexpensive, safe, and effective method to improve healing and prevent hypertrophic scarring in resource-limited settings, potentially changing standard practice for donor site management.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age 2 years and above, of any gender.

Patients requiring a split-thickness skin graft.

Patients giving informed consent for study participation.

Patients with serum albumin > 3 g/dL.

Exclusion Criteria:

* Patients allergic to heparin.

Patients with diabetes, hematological disorders, kidney or liver diseases, or malignancies.

Patients on medications affecting wound healing.

Patients with existing hypertrophic scarring at the donor site

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-09-10 (Actual)

PRIMARY OUTCOMES:
Incidence of hypertrophic scarring at STSG donor site | Assessed at 10th post-operative day, 1 month, and 3 months
  Hypertrophic scarring will be measured using the Vancouver Scar Scale, which evaluates vascularity, height, pliability, and pigmentation. Total score ranges from 0-13. Comparison will be made between the standard dressing and heparin dressing groups.

SECONDARY OUTCOMES:
Donor site pain | 10th post-operative day, 1 month, and 3 months
  Pain will be assessed using the Numeric Rating Scale (0-10), where 0 indicates no pain and 10 indicates worst pain. Daily analgesic requirement will also be documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Plastic & Reconstructive Surgery Department, Ruth Pfau Civil Hospita, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No